CLINICAL TRIAL: NCT06163352
Title: The Effect of Vasopressor Agents on Pressure Injury Development in Intensive Care Patients
Brief Title: The Effect of Vasopressor on Pressure Injury Development
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Koç University (Other)
Responsible Party: Principal Investigator, Ayda Kebapci, Associate Professor, Koç University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: PU
Record Dates: First submitted 2023-11-14; First posted 2023-12-08 (Actual); Last update posted 2023-12-21 (Actual); Status verified 2023-12

CONDITIONS: Vasopressor Adverse Reaction; Pressure Injury; Pressure Ulcer
Keywords: vasopressor; pressure injury; pressure ulcer; development risk; prevention
MeSH Terms: conditions — Pressure Ulcer | interventions — Norepinephrine; Dopamine

STUDY DESIGN:
Intervention Model Description: Patients with pressure injury (n=64) and patients without pressure injury (n=84)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients with pressure injury (Experimental): The intervention is vasopressor infusion. In this am, 64 surgical and medical patients treated with vasopressor agents in the intensive care unit and developed pressure injury were included.
  Interventions: Drug: Norepinephrine
- Patients without pressure injury (Active Comparator): The intervention is vasopressor infusion. In this arm, 84 surgical and medical patients treated with vasopressor agents in the intensive care unit and did not develop pressure injury were included.
  Interventions: Drug: Norepinephrine

INTERVENTIONS:
Drug: Norepinephrine — The sample consisted of all medical and surgical patients over 18 who do not have pressure injury upon admission and received one or more vasopressor agent infusions (norepinephrine, epinephrine, dopamine) for at least 48 hours during their stay in the ICU and pressure injury development was assessed. The effect of combined use of more than one vasopressor agent on the development of pressure injury was investigated, considering the type and quantity of vasopressors (norepinephrine and dopamine), vasopressor combinations, total duration of infusion, and doses of vasopressors used.
  Other Names: dopamine

SUMMARY:
Background: Vasopressors are life-saving agents that increase mean arterial pressure. The pharmacodynamic features of these agents and previous studies suggest that vasopressors may be an essential risk factor in developing pressure injuries.

Objective: This study aimed to examine the effect of vasopressors in medical-surgical intensive care patients on pressure injury development.

Design and Settings: This retrospective and correlational study was conducted between March 2021- May 2022. The electronic patient data were obtained from 148 surgical and medical patients treated with vasopressor agents in the intensive care unit. Data on patients' demographic and clinical characteristics were evaluated using descriptive statistical methods (number, percentage, mean, standard deviation). A logistic regression model was established to estimate the dependent variable (development of pressure injury) with the independent variables.

DETAILED DESCRIPTION:
There is a need for studies in which vasopressor drugs are discussed in detail and the risk factors that may cause pressure injury development in patients. Therefore, this study aims to examine vasopressors' effect on PI development among patients in intensive care units.

MATERIALS and METHODS Design This retrospective and correlational study examined the effect of vasopressors on pressure injury development in medical and surgical intensive care patients. The Consolidated Standards of Reporting Trials (CONSORT) statement guided this study (Boutron et al. , 2008) Ethics Approval The Ethics Committee of Koç University approved the study (2022.365.IRB1.155), and institutional permission was obtained.

Sample and Settings The study included all medical-surgical adult critical patients hospitalized in the 16-bed Adult Intensive Care Unit (ICU). It is a 3rd level ICU where medical and surgical patients receive life support treatments and care at the highest level. The study was conducted at XXX Hospital between May 2020 and March 2021. The study population consisted of 900 patients hospitalized in the ICU between these dates. The sample consisted of all medical and surgical patients over 18 who do not have pressure injury upon admission and received one or more vasopressor agent infusions (norepinephrine, epinephrine, phenylephrine, dopamine, adrenaline, dobutamine) for at least 48 hours during their stay in the ICU. Nurses checked skin and the existence of PI daily. They recorded their findings during the stay of the patients in the Pressure Wound Prevention Evaluation and Follow-up Form within 24 hours. Prevention, diagnosis, staging of pressure injury, and implementation of interventions appropriate to the stage were performed per this protocol. If pressure injury develops in patients, it is evaluated and staged, and appropriate interventions are decided for each patient under the leadership of the wound care nurse. After the first evaluation of the PI by the wound care nurse, the wound care nurse continued to evaluate patients' wounds daily. In line with all these approaches, it aimed to provide standardization for managing pressure injury prevention, staging, and implementation of interventions and to provide the highest reliability between nurses' evaluations and interventions. In line with this protocol, In the ICU, barrier cream or spray and gel adhesive dressings were used on the pressure areas of the body parts for prevention, and support skin surfaces were used to distribute the pressure by the pressure injury protocol.

Furthermore, skin hygiene and nourishing, applying gel adhesive dressing on pressure areas, repositioning of sedated patients every 2 hours, frequent position changes of unsedated patients, heel and head elevation, and nutritional assessment of patients were implemented to prevent PI. The European Pressure Ulcer Advisory Panel and the National Pressure Ulcer Advisory Panel Pressure Ulcers Classification System used by the nurses to stage the pressure injury of the accordingly Stage I (Nonblanchable erythema of intact skin), stage II (Partial-thickness skin loss with exposed dermis), stage III (Full-thickness skin loss), stage IV (Full-thickness skin and tissue loss), unstageable stage (Obscured full-thickness skin and tissue loss), and suspected deep tissue injury (Persistent nonblanchable deep red, maroon, or purple discoloration) (Edsberg, Black, 2016). All nurses working in the ICU attended the orientation training program before starting to work in the ICU and received formal training on pressure injury prevention, diagnosis, staging, and planning and implementation of appropriate interventions within the scope of this program.

Data Collection Data were obtained retrospectively from the electronic health record system by the researchers. The authors developed a data collection form to collect data. Data regarding the demographic characteristics included sex, age, and comorbid diseases. Clinical data included the diagnosis for ICU admission (medical/surgical), mechanical ventilation (MV) requirement and duration of MV, the total length of stay in ICU, the types of vasopressors used, the mean daily dose, and the duration of infusion of the vasopressor agents were recorded. The other PI risk factors (age>65, receiving chemotherapy, cachexia, being at the end of life, circulation problems, dehydration, and loss of sensation) were also determined. The data regarding the PI were obtained from the Pressure Wound Evaluation and Follow-up Form used by ICU nurses. Furthermore, the location, stage (based on the National Pressure Injury Advisory Panel staging system), and the time for PI development were between initiation of vasopressor vasopressor and pressure injury. In the case of PI development in patients, PI was staged under the leadership of the wound care nurse to provide standardization for pressure injury prevention, diagnosis staging, and the implementation of appropriate interventions in all patients.

Statistical Analysis Data was analyzed using SPSS (Statistical Package for Social Sciences) for Windows 28.0 program (IBM Corp.; Armonk, NY, USA). Data on patients' demographic and clinical characteristics were evaluated using descriptive statistical methods (number, percentage, mean, standard deviation). A logistic regression model was established to estimate the dependent variable (development of PI) with the independent variables. The significance was evaluated at p<.05. Only statistically significant variables found at the 0.05 level were included in the model table; the statistically unsignificant variables were removed from the model, and the final model was decided. Using the logistic regression model and if the R2 value is 58.9%, the minimum number of samples was 97% at the 95% confidence 95% power level, and 5% standard error. Therefore, 148 participants were enough for regression analysis.

ELIGIBILITY:
Inclusion Criteria:

The sample consisted of all:

* Medical and surgical patients over 18 who do not have pressure injury upon admission
* Received one or more vasopressor agent infusions (norepinephrine, epinephrine, phenylephrine, dopamine, adrenaline, dobutamine) for at least 48 hours during their stay in the intensive care unit

Exclusion Criteria:

* patients less than 18 years old
* less than 48 hours stay in intensive care unit
* did not receive ant vasospressor agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 148 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2023-08-01 (Actual); Study Completion 2023-09-01 (Actual)

PRIMARY OUTCOMES:
Development of pressure injury | 14 months
  The development of the pressure injury was followed and the data regarding the PI were obtained from the Pressure Wound Evaluation and Follow-up Form.

CONTACTS AND LOCATIONS:
Overall Officials: Ayda Kebapci, Assoc Prof, Principal Investigator — Koç University
Locations (1):
- Koç University, Istanbul, None Selected, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tayyib N, Coyer F, Lewis P. Saudi Arabian adult intensive care unit pressure ulcer incidence and risk factors: a prospective cohort study. Int Wound J. 2016 Oct;13(5):912-9. doi: 10.1111/iwj.12406. Epub 2015 Feb 9. PMID 25662591
- [Background] Tschannen D, Bates O, Talsma A, Guo Y. Patient-specific and surgical characteristics in the development of pressure ulcers. Am J Crit Care. 2012 Mar;21(2):116-25. doi: 10.4037/ajcc2012716. PMID 22381988
- [Background] European Pressure Ulcer Advisory Panel (EPUAP), National Pressure Injury Advisory Panel (NPUAP) and Pan Pacific Pressure Injury Alliance (2019). Prevention and Treatment of Pressure Ulcers/Injuries: Quick Reference Guide. Emily Haesler (Ed.). https://static1.squarespace.com/static/6479484083027f25a6246fcb/t/647dc6c178b260694b5c9365/1685964483662/Quick_Reference_Guide-10Mar2019.pdf (accessed: 11/13/2023).
- [Background] Lima Serrano M, Gonzalez Mendez MI, Carrasco Cebollero FM, Lima Rodriguez JS. Risk factors for pressure ulcer development in Intensive Care Units: A systematic review. Med Intensiva. 2017 Aug-Sep;41(6):339-346. doi: 10.1016/j.medin.2016.09.003. Epub 2016 Oct 22. English, Spanish. PMID 27780589
- [Background] Oczkowski S, Alshamsi F, Belley-Cote E, Centofanti JE, Hylander Moller M, Nunnaly ME, Alhazzani W. Surviving Sepsis Campaign Guidelines 2021: highlights for the practicing clinician. Pol Arch Intern Med. 2022 Aug 22;132(7-8):16290. doi: 10.20452/pamw.16290. Epub 2022 Jul 6. PMID 35791800
- [Background] Nijs N, Toppets A, Defloor T, Bernaerts K, Milisen K, Van Den Berghe G. Incidence and risk factors for pressure ulcers in the intensive care unit. J Clin Nurs. 2009 May;18(9):1258-66. doi: 10.1111/j.1365-2702.2008.02554.x. Epub 2008 Dec 11. PMID 19077028
- [Background] Cox J, Roche S, Murphy V. Pressure Injury Risk Factors in Critical Care Patients: A Descriptive Analysis. Adv Skin Wound Care. 2018 Jul;31(7):328-334. doi: 10.1097/01.ASW.0000534699.50162.4e. PMID 29923903
- [Background] Edsberg LE, Black JM, Goldberg M, McNichol L, Moore L, Sieggreen M. Revised National Pressure Ulcer Advisory Panel Pressure Injury Staging System: Revised Pressure Injury Staging System. J Wound Ostomy Continence Nurs. 2016 Nov/Dec;43(6):585-597. doi: 10.1097/WON.0000000000000281. PMID 27749790
- [Derived] Kebapci A, Tilki R. The effect of vasopressor agents on pressure injury development in intensive care patients. Intensive Crit Care Nurs. 2024 Aug;83:103630. doi: 10.1016/j.iccn.2024.103630. Epub 2024 Mar 12. PMID 38479195